CLINICAL TRIAL: NCT05407805
Title: A LOW-INTERVENTIONAL LONGITUDINAL STUDY OF AN ELECTRONIC SICKLE CELL DISEASE PATIENT REPORTED OUTCOMES IN ADULT PARTICIPANTS AGED ≥18 YEARS OF AGE ON AND OFF HYDROXYUREA
Brief Title: A Study to Learn About Sickle Cell Disease In Adult Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4071008
Record Dates: First submitted 2022-05-18; First posted 2022-06-07 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Sickle Cell Disease
Keywords: Vaso-occlusive crisis (VOC); Hemoglobin S (HbS)
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Sickle Cell Trait

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Control Group: SCD participants not on disease modifying treatment.
  Interventions: Other: Electronic Diary
- SCD Disease Modifying Treatment Group: SCD participants on a stable dose of a SCD disease modifying treatment regimen.
  Interventions: Other: Electronic Diary

INTERVENTIONS:
Other: Electronic Diary — Participants will be asked to complete a daily electronic patient reported outcome diary entry to report on their experience in the past 24 hours.
  Other Names: SCD electronic patient reported outcome (ePRO)

SUMMARY:
The purpose of this clinical trial is to evaluate the performance of the sickle cell disease (SCD) electronic diary in people with SCD who are on treatment that will change SCD and those not on such a treatment.

SCD is a type of condition when there are fewer red blood cells to carry oxygen around the body.

This disease can be passed on from parent to child and may cause pain, infections and damage to organs.

This study is seeking participants who:

* are confirmed with SCD
* are on a stable regimen of disease changing treatment or have not received any disease changing treatment before the start of the study and do not plan any changes in their treatment during the 6-month study observation period For 6 months, participants will be asked to complete a daily electronic diary to report on their experience in the past 24 hours with sickle cell pain crisis (if they got any treatment and what medications they took), worst pain, worst tiredness, and their ability to perform usual physical activities. We will compare the experiences of people who are taking SCD-modifying therapy to those that are not taking a SCD-modifying therapy.

ELIGIBILITY:
Inclusion Criteria (All Groups):

- Confirmed diagnosis of stable SCD (HbS/S or HbS/beta-zero-thalassemia).

Additional Inclusion Criteria (No Disease Modifying Treatment Control Group):

* Have experienced ≥1 episode(s) of medical utilization (MU) VOC within 12 months prior to Screening.
* Data available for number of MU VOC(s) during the 12-month interval prior to Screening and a value for %fetal hemoglobin (HbF) collected subsequent to 1 year of age in the absence of recent transfusion.

Additional Inclusion Criteria (SCD Disease Modifying Treatment Group):

* Have experienced ≥1 episode(s) of MU VOC within 12 months prior to initiation of HU and/or crizanlizumab (whichever was initiated earlier).
* Must be on a stable dose of their SCD treatment regimen ≥8 weeks prior to Day 1 with the intent of remaining on the same dose throughout the study, unless adjustments are medically necessary due to bone marrow suppression, in accordance with published guidelines and/or product specific guidance (eg, package label). Accepted SCD disease modifying treatment regimens include:

  * HU alone and/or in combination with crizanlizumab, L-glutamine and/or voxelotor; or
  * Crizanlizumab alone and/or in combination with HU, L-glutamine and/or voxelotor.
* Data available for number of MU VOC(s) during the 12-month interval prior to initiation of any SCD disease modifying treatment, as described above, and a value for %HbF collected subsequent to 1 year of age, prior to initiation of any HU treatment, and in the absence of recent transfusion.

Exclusion Criteria (All Groups):

* Evidence or history of ongoing (condition or sequelae) clinically significant hematological (non-SCD), renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including overt stroke but excluding silent cerebral infarct), hepatic (excluding cholelithiasis), psychiatric or neurological disease as assessed from medical records.
* Marked ongoing bone marrow suppression as evidenced by any of the following as per medical record: severe anemia, absolute neutrophil count (ANC) <1000 mm3 white blood cell (WBC), thrombocytopenia (platelet count <100,000 mm3) within ≤8 weeks prior to Day 1 enrollment.
* History of hematopoietic stem cell transplant or treatment with gene therapy as assessed from medical records.
* History of simple transfusion within ≤4 weeks prior to Day 1 enrollment as assessed from medical records or participant self-report.
* History of chronic transfusion/exchange transfusion within ≤12 weeks prior to Day 1 enrollment as assessed from medical records or participant self-report and/or plan to initiate such treatment during the 6-month observation period.

Additional Exclusion Criteria (No Disease Modifying Treatment Control Group):

* Participant received HU and/or crizanlizumab at any time within ≤18 months of Day 1 enrollment and treatment(s) was discontinued due to lack of efficacy (no reduction in the frequency of VOCs, documented or perceived) and/or plan to initiate said treatment(s) during the 6-month observation period.
* Participant received voxelotor or L-glutamine within ≤4 weeks of Day 1 enrollment and/or plan to initiate said treatment(s) during the 6-month observation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a confirmed diagnosis of stable Sickle Cell Disease (SCD) (hemoglobin S inherited from both parents [HbS/S] or hemoglobin S inherited from one parent and hemoglobin beta thalassemia inherited from the other parent [HbS/beta-zero-thalassemia] genotype) who are either not on disease modifying treatment or on a stable dose of a SCD disease modifying treatment regimen.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Physician-reported Medical Utilization vaso-occlusive crisis (VOC) rate | Day 1 to 180
  Confirmation that the population is suitable for assessing responsiveness of electronic patient reported outcomes based upon a lower frequency rate of Physician reported Medical Utilization VOCs in the SCD disease modifying treatment group.
VOC Day rate | Day 1 to 180
  Responsiveness of electronic patient reported outcomes between participants treated with SCD disease modifying treatment or no disease modifying treatment.
Patient-reported VOC Event rate | Day 1 to 180
  Responsiveness of electronic patient reported outcomes between participants treated with SCD disease modifying treatment or no disease modifying treatment.
Average SCD ePRO daily worst pain score during VOC days | Day 1 to 180
  Responsiveness of electronic patient reported outcomes between participants treated with SCD disease modifying treatment or no disease modifying treatment.
Average SCD ePRO daily worst pain score during non-VOC days | Day 1 to 180
  Responsiveness of electronic patient reported outcomes between participants treated with SCD disease modifying treatment or no disease modifying treatment.
Average SCD ePRO daily worst tiredness score during VOC days | Day 1 to 180
  Responsiveness of electronic patient reported outcomes between participants treated with SCD disease modifying treatment or no disease modifying treatment.
Average SCD ePRO daily worst tiredness score during non-VOC days | Day 1 to 180
  Responsiveness of electronic patient reported outcomes between participants treated with SCD disease modifying treatment or no disease modifying treatment.
Average SCD ePRO daily rating for ability to perform usual physical activity during a VOC day | Day 1 to 180
  Responsiveness of electronic patient reported outcomes between participants treated with SCD disease modifying treatment or no disease modifying treatment.
Average SCD ePRO daily rating for ability to perform usual physical activity during a non-VOC day | Day 1 to 180
  Responsiveness of electronic patient reported outcomes between participants treated with SCD disease modifying treatment or no disease modifying treatment.

SECONDARY OUTCOMES:
Quantitative relationship between VOC Day rate and Physician-reported Medical Utilization VOC | Day 1 to 180
  Quantitative measure of association between VOC Day rate and Physician-reported Medical Utilization VOC.
Quantitative relationship between VOC Day rate and Physician-reported Medical Utilization VOC rate across treatment groups | Day 1 to 180
  Comparison of quantitative measures of treatment effect between VOC Day rate and Physician-reported Medical Utilization VOC rate.
Quantitative relationship between Patient-reported VOC Event rate and Physician-reported Medical Utilization VOC rate | Day 1 to 180
  Quantitative measure of association between Patient-reported VOC Event rate and Physician-reported Medical Utilization VOC rate.
Quantitative relationship between Patient-reported VOC Event rate and Physician-reported Medical Utilization VOC rate across treatment groups | Day 1 to 180
  Comparison of quantitative measures of treatment effect between Patient-reported VOC Event rate and Physician-reported Medical Utilization VOC rate.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Foundation for Sickle Cell Disease Research, Hollywood, Florida
  - Mid-Atlantic Permanente Medical Group Largo Medical Center, Largo, Maryland
  - Mid-Atlantic Permanente Medical Group Largo Medical Center, Upper Marlboro, Maryland
  - Sanguine Biosciences, Inc., Waltham, Massachusetts
  - Cohen Children's Medical Center, New Hyde Park, New York

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4071008